CLINICAL TRIAL: NCT04892823
Title: Accelerated Biological and Phenotypic Aging in Hematopoietic Cell Transplant Survivors: Social Support as a Protective Factor
Brief Title: Social Relationships and Accelerated Aging in Hematopoietic Cell Transplant Survivors
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kelly E Rentscher, PhD, Principal Investigator, Medical College of Wisconsin
Other Study IDs: 43000; NCI-2021-02616 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 43000 (Other: Medical College of Wisconsin); K01AG065485 (NIH)
Record Dates: First submitted 2021-05-10; First posted 2021-05-19 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Supportive care (EAR, questionnaires, biospecimen collection): Participants will complete comprehensive assessments of social processes at 100 days and 1 year after HCT that combine reports of social support, strain, and isolation with a naturalistic observation tool, the Electronically Activated Recorder (EAR), which captures ambient sound bites to assess social interactions in survivors' daily lives. At each time point, participants will also provide reports of symptoms to characterize phenotypic aging, including cognitive, physical, and functional complaints, and blood samples to assess biological aging, including cellular senescence, DNA damage, SASP, and cellular stress using genome wide RNA sequencing. Relevant clinical information that could influence biological aging will also be collected from patients' medical records to consider as covariates.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood sample
Other: Electronic Health Record Review — Review of medical records
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This project aims to elucidate the important protective elements of social relationships and identify concrete, modifiable behavioral factors that contribute to biological and phenotypic aging in hematopoietic cell transplantation (HCT) survivors and can be used to develop biologically informed interventions to improve quality of life and prolong the healthspan of individuals with accelerated aging.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine associations between social support, strain, and isolation and phenotypic aging over the 1-year recovery period.

II. Examine associations between social support, strain, and isolation and biological aging over the 1-year recovery period.

III. Test biological aging as a mediator linking social processes and phenotypic aging.

EXPLORATORY OBJECTIVE:

I. Test sex differences in Aims 1 and 2.

OUTLINE:

Adopting a prospective design, participants will complete comprehensive assessments of social processes at 100 days and 1 year after HCT that combine reports of social support, strain, and isolation with a naturalistic observation tool, the Electronically Activated Recorder (EAR), which captures ambient sound bites to assess social interactions in survivors' daily lives16. At each time point, participants will also provide reports of symptoms to characterize phenotypic aging, including cognitive, physical, and functional complaints, and blood samples to assess biological aging, including cellular senescence, DNA damage, SASP, and cellular stress using genome-wide RNA sequencing. Relevant clinical information that could influence biological aging will also be collected from patients' medical records to consider as covariates.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older who are competent to give their informed consent.
* Ability to read, speak, and understand English.
* Received a hematopoietic cell transplant within the previous 100 days.

Exclusion Criteria:

* Less then Aged 18 years and older who are competent to give their informed consent.
* Cannot read, speak, and understand English.
* Has not received a hematopoietic cell transplant within the previous 100 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing HCT for hematologic cancers.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The number of participants with gene expression of cellular senescence marker p16. | Day 100 and 1 year post-transplant
  This will be measured by mRNA/gene expression.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Rentscher, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No